CLINICAL TRIAL: NCT05918705
Title: Is the Ratio of Optic Nerve Sheath Diameter to Eyeball Transverse Diameter Correlated with the Prognosis of Sepsis Associated Encephalopathy in Critically Ill Patients
Brief Title: Optic Nerve Sheath Diameter / Eyeball Transverse Diameter Ratio and Prognosis of Sepsis Associated Encephalopathy
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Ashraf Torki, Lecturer of Anesthesia, Zagazig University (Principal Investigator), Zagazig University
Other Study IDs: ZU-IRB #10413
Record Dates: First submitted 2023-06-05; First posted 2023-06-26 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Sepsis-associated Encephalopathy
Keywords: Optic nerve sheath diameter; Eyeball transverse diameter; Sepsis-associated encephalopathy
MeSH Terms: conditions — Sepsis-Associated Encephalopathy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- ONSD / ETD Ratio Correlation With Prognosis of Sepsis Associated Encephalopathy: * Data on in-hospital mortality will be recorded for all patients.
  * Clinical diagnosis of brain death will be also recorded for all patients.
  * Morbidity will be assessed both on ICU discharge and 3 months following ICU discharge with the Modified Rankin Scale (mRS), where patients will be assessed at the 3-month follow-up by telephone or face-to-face interviews with the patients or relatives.
  According to neurologic outcome on ICU discharge and 3 months following ICU discharge, the included patients will be classified into two groups;
  * Good Neurologic Outcome (GNO); mRS 0 - 2.
  * Poor Neurologic Outcome (PNO); mRS 3 - 6.
  Interventions: Procedure: Ultrasound optic nerve sheath diameter / eyeball transverse diameter ratio

INTERVENTIONS:
Procedure: Ultrasound optic nerve sheath diameter / eyeball transverse diameter ratio — Ocular ultrasonography will be performed once daily on patients diagnosed with sepsis associated encephalopathy at the bedside by two experienced examiners, who will be blinded to patients' clinical data, following the CLOSED protocol for ONSD sonography.
  ONSD will be measured at 3 mm behind the merging point of the nerve from the papilla "optic disc". The maximum external diameter of ONSD will be measured in the transverse plane perpendicular to the optic nerve and the maximum diameter of ETD (parallel lens) on this plane will be measured.
  Two measurements will be taken for each eye; horizontal and vertical. The sequence for measurements will be left eye horizontal; left eye vertical; right eye horizontal; right eye vertical.
  The ONSD measurements in the transversal and the sagittal plane for each eye measured by the two examiners will be averaged. Then, ETDs measurements will be averaged to obtain averaged ONSD/ETD ratio as a data to record the mean values of ONSD/ETD ratio.

SUMMARY:
Sepsis is associated with a mortality rate of 20-25%, with significant increase in case of associated comorbidities or shock. SAE is one of the most common forms of encephalopathy encountered in critically ill patients, with increased ICP as a possible underlying mechanism. Many studies revealed that ONSD is a valuable ICP monitoring tool. Also, ONSD/ETD ratio, according to previous studies, seemed to be more reliable than ONSD alone in predicting neurological outcomes of comatosed patients. The present study will assess the correlation between US-ONSD/ETD ratio and the prognosis of SAE in critically ill patients.

DETAILED DESCRIPTION:
Site of the Study: Surgical intensive care units, Zagazig University Hospitals.

Duration of Study: Around 6 months. Type of the Study: Prospective observational study.

Sample Size:

Sample size is calculated to be 89 patients assuming that the area under curve (AUC) of the ONSD/ETD ratio in predicting prognosis of comatose patients was 0.808 (95%CI: 0.696 - 0.920) with confidence level 0.95.

Withdrawal Criteria:

The patient has the right to withdraw from the study at any time without any negative consequences on treatment plan.

The following cases also will be withdrawn from the study;

* Cases diagnosed with toxic or metabolic encephalopathy.
* Cases with failed US-ONSD measurement due to unclear US images.
* Cases transferred to another hospital during treatment course. ii- study design: All patients will undergo head CT scan on the first day of disturbed conscious level onset for etiology assessment to exclude intracranial pathology.

Informed written consent will be obtained from one of patient's 1st degree relatives due to patient's disturbed conscious level.

Patient Assessment:

All patients will be assessed by meticulous history taking, clinical examination, and standard laboratory workup. Critically ill patients diagnosed with SAE, sedated or unconscious, and on invasive mechanical ventilation will be enrolled in our study. The severity of clinical illness will be assessed using the acute physiology and chronic health evaluation II (APACHE II) on ICU admission. Sequential organ failure assessment (SOFA) score will be used to assess the incidence of organ dysfunction/failure due to sepsis and will be calculated daily.

Patients will be followed up till either in-hospital mortality or hospital discharge. Discharged patients will be then followed up till 3 months follow-up by telephone or face-to-face interviews with the patients or relatives for morbidity assessment.

Measurement of US Ratio of ONSD/ETD Ocular ultrasonography will be performed once daily at the bedside by two experienced examiners, who will be blinded to patients' clinical data, following the CLOSED protocol for ONSD sonography;

* Color Doppler; to identify central retinal artery (CRA), central retinal vein (CRV), and ophthalmic artery (OA) to better detect optic nerve course.
* Low power output; the retina, a sensitive organ, requires the lowest possible output power for a safe use of diagnostic US.
* Optic disk clarity; the clearance of the optic disk is a minimum requirement for a correct landmark 3 mm behind the papilla.
* Safety (short examination duration); minimize image information loss recording an US video clip to reduce the examination duration for the safety of the patient (ALARA principle "as low as reasonable achievable")
* Elevate frequency; for a better quality of US images.
* Dual measurements; two measurements should be taken for each eye: horizontal and vertical.

US Machine Setup:

The liner high frequency probe 7 - 12 MHz of SonoSite M-Turbo ultrasound machine will be used. Power will be reduced to achieve a mechanical Index (MI) ≤ 0.23 and frequency will be kept at 10 MHz "ALARA principle" to safeguard the patient's eye from possible potential biological damage.

Positioning:

* The patient will be supine in neutral head position with the eyelids closed.
* The operator will sit behind the patient's head. Care will be taken so that probe-cable will not be in tension or suspension, in order to minimize tension, which limits fine movements. The operator hand holding the probe will rest on the patient's forehead, to prevent unnecessary pressure being exerted on the eye. Pressure with the probe on the eyeball will be also minimized.

Preparation:

Tegaderm will be placed on the closed eyelid to prevent possible direct contact between the eye and the gel. A layer of US gel will be applied to avoid air between probe and skin.

US Scanning:

During horizontal measurement, the probe will be placed at an approximate angle of 15°-20° on the patient's closed upper eyelid. For the vertical measurement, the probe should be placed on the center of the patient's closed eye, slightly toward the corner of the nose (latero-to-medial direction), trying to intercept the nerve direction.

The probe will be placed horizontally above the transverse axis of the eyeball and then slowly and vertically moved to the eyeball from the patient's forehead to the nose until the clearest and artifact-free optimal plane was echoed on the frozen images. The optic nerve image was a low-echo strip structure located in the front and rear of the eyeball. The simultaneous appearance of lens and optic nerve meant the US probe was on the best plane. After removing the probe, the optic nerve and the sheaths on its two sides were visible with distinct margins.

- Color Doppler: According to the CLOSED protocol, the use of color Doppler is mandatory to minimize errors induced by acoustic shadow cones and false images due to inadequate quality of B-mode. Color Doppler will visualize CRA and CRV, which run in the middle of the distal segment of the ON. CRA and CRV visualization will aid to correctly identify the ON course, which can be difficult due to artifacts, wrong angulation of the probe, and nerve tortuosity. Thus, these vessels will be used as landmarks to identify the correct anatomical plane for reliable ONSD measurements. If needed, color Doppler also will visualize OA, which runs parallel to the ON, for more accurate identification of ONSD margins.

ONSD Measurement:

ONSD will be measured at 3 mm behind the merging point of the nerve from the papilla "optic disc", since at this distance, the sheath is subject to maximum diameter fluctuations due to ICP (the point of greatest distensibility). The maximum external diameter of ONSD will be measured in the transverse plane perpendicular to the optic nerve and the maximum diameter of ETD (parallel lens) on this plane will be measured.

Two measurements (dual measurements) will be taken for each eye; horizontal and vertical. The best captured frame will be used for measurements to minimize any operator-dependent error. In case of doubt or clear discrepancies between the horizontal and vertical measurements, the horizontal measure will be considered as most reliable. The sequence for measurements will be left eye horizontal; left eye vertical; right eye horizontal; right eye vertical. To reduce the examination time, we will capture a short video clip, from which the performer can then extract the best frame for measurement.

The ONSD measurements in the transversal and the sagittal plane for each eye measured by the two examiners will be averaged. Then, ETDs measurements will be averaged to obtain averaged ONSD/ETD ratio as a data to record the mean values of ONSD/ETD ratio.

Measured Data:

1. Demographic data including age, sex, body mass index (BMI).
2. Patients' comorbidities.
3. Averaged ONSD/ETD ratio; measured once daily until ICU discharge or death.
4. Vital signs; including mean blood pressure (MAP) and heart rate (HR) at time of ONSD/ETD measurement.
5. Need for vasopressor and/or inotropic support at time of ONSD/ETD measurement.
6. ICU day for ONSD/ETD measurement.
7. Ratio of PaO2/FiO2 (PFI), PaCO2 at time of ONSD/ETD measurement.
8. Occurrence of acute kidney injury (AKI) at time of ONSD/ETD measurement.
9. PEEP, peak airway pressure, pressure support/pressure control setting and ventilator mode at time of ONSD/ETD measurement.
10. ICU- length of stay (ICU-LOS), 90-day mortality and number of days alive during the first 90 days from admission to the ICU, from electronic patient charts.

Measured Scores:

1. APACHE II score on ICU admission.
2. SOFA score daily.
3. Full Outline of UnResponsiveness (FOUR) score at time of ONSD/ETD measurement.
4. Modified Rankin Scale (mRS) for Neurological Outcome:

   * Data on in-hospital mortality will be recorded for all patients.
   * Clinical diagnosis of brain death will be also recorded for all patients.
   * Morbidity will be assessed both on ICU discharge and 3 months following ICU discharge with the Modified Rankin Scale (mRS), where patients will be assessed at the 3-month follow-up by telephone or face-to-face interviews with the patients or relatives.

According to neurologic outcome on ICU discharge and 3 months following ICU discharge, the included patients will be classified into two groups; Good Neurologic Outcome (GNO); mRS 0 - 2. Poor Neurologic Outcome (PNO); mRS 3 - 6.

ELIGIBILITY:
Inclusion Criteria:

1. Acceptance of one of patient's 1st degree relatives.
2. Age ≥ 18 and ≤ 65 years old of both sexes.
3. Sedated or unconscious patients and on invasive mechanical ventilation.
4. Patients diagnosed with sepsis associated encephalopathy (SAE);

Exclusion Criteria:

1. Ocular and/or optic nerve pathology; e.g., ocular trauma or surgery, previous ocular pathology as glaucoma or cataract, conjunctival or orbital edema, vitreous hemorrhage and optic nerve disease or injury.
2. Intracranial pathology; e.g., central nervous system (CNS) infection, cerebrovascular accident, cerebral hemorrhage, brain trauma or tumor, and any previous neurosurgical procedure.
3. Toxic or metabolic encephalopathy, e.g., alcohol toxicity, liver or kidney disease.
4. Serious co-morbidities that could affect life expectancy, e.g., hematopathy or cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SAE will be diagnosed by the combination of extracranial infection and clinical signs of neurological dysfunction. SAE clinical manifestations include impairment of awareness, which ranges from delirium to coma.
Sampling Method: Probability Sample
Enrollment: 89 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-10 (Actual)

PRIMARY OUTCOMES:
Correlation between US ratio of ONSD/ETD and neurologic outcome 3 months following ICU discharge in critically ill patients with SAE. | 3 months following ICU discharge
  Correlation between US ratio of ONSD/ETD and neurologic outcome 3 months following ICU discharge in critically ill patients with SAE.

SECONDARY OUTCOMES:
Correlation between US ratio of ONSD/ETD and neurologic outcome on ICU discharge in critically ill patients with SAE. | From date of enrolling in the study until the date of discharge from ICU or date of death from any cause, whichever came first, assessed up to 90-days
  Correlation between US ratio of ONSD/ETD and neurologic outcome on ICU discharge in critically ill patients with SAE.
Correlation between US ratio of ONSD/ETD and 90-day mortality in critically ill patients with SAE. | 90-days
  Correlation between US ratio of ONSD/ETD and 90-day mortality in critically ill patients with SAE.
Correlation between US ratio of ONSD/ETD and ICU-LOS in critically ill patients with SAE. | From date of enrolling in the study until the date of discharge from ICU or date of death from any cause, whichever came first, assessed up to 90-days
  Correlation between US ratio of ONSD/ETD and ICU-LOS in critically ill patients with SAE.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf Torki, MD, Principal Investigator — Anesthesia and surgical intensive care, zagazig university, faculty of medicine; Mona Shahin, MD, Study Director — Anesthesia and surgical intensive care, zagazig university, faculty of medicine; Sherif MS Mowafy, MD, Study Director — Anesthesia and surgical intensive care, zagazig university, faculty of medicine
Locations (1):
- Ashraf Torki, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Raffiz M, Abdullah JM. Optic nerve sheath diameter measurement: a means of detecting raised ICP in adult traumatic and non-traumatic neurosurgical patients. Am J Emerg Med. 2017 Jan;35(1):150-153. doi: 10.1016/j.ajem.2016.09.044. Epub 2016 Sep 23. PMID 27852525
- [Background] Zhu S, Cheng C, Zhao D, Zhao Y, Liu X, Zhang J. The clinical and prognostic values of optic nerve sheath diameter and optic nerve sheath diameter/eyeball transverse diameter ratio in comatose patients with supratentorial lesions. BMC Neurol. 2021 Jul 2;21(1):259. doi: 10.1186/s12883-021-02285-7. PMID 34215217
- [Background] Onder H, Goksungur G, Eliacik S, Ulusoy EK, Arslan G. The significance of ONSD, ONSD/ETD ratio, and other neuroimaging parameters in idiopathic intracranial hypertension. Neurol Res. 2021 Dec;43(12):1098-1106. doi: 10.1080/01616412.2021.1949688. Epub 2021 Aug 19. PMID 34409925
- [Background] Hassen GW, Bruck I, Donahue J, Mason B, Sweeney B, Saab W, Weedon J, Patel N, Perry K, Matari H, Jaiswal R, Kalantari H. Accuracy of optic nerve sheath diameter measurement by emergency physicians using bedside ultrasound. J Emerg Med. 2015 Apr;48(4):450-7. doi: 10.1016/j.jemermed.2014.09.060. Epub 2014 Dec 9. PMID 25497897
- [Background] Zhu S, Cheng C, Wang LL, Zhao DJ, Zhao YL, Liu XZ. Prognostic values of optic nerve sheath diameter for comatose patients with acute stroke: An observational study. World J Clin Cases. 2022 Nov 26;10(33):12175-12183. doi: 10.12998/wjcc.v10.i33.12175. PMID 36483822
- [Background] Rhodes A, Evans LE, Alhazzani W, Levy MM, Antonelli M, Ferrer R, Kumar A, Sevransky JE, Sprung CL, Nunnally ME, Rochwerg B, Rubenfeld GD, Angus DC, Annane D, Beale RJ, Bellinghan GJ, Bernard GR, Chiche JD, Coopersmith C, De Backer DP, French CJ, Fujishima S, Gerlach H, Hidalgo JL, Hollenberg SM, Jones AE, Karnad DR, Kleinpell RM, Koh Y, Lisboa TC, Machado FR, Marini JJ, Marshall JC, Mazuski JE, McIntyre LA, McLean AS, Mehta S, Moreno RP, Myburgh J, Navalesi P, Nishida O, Osborn TM, Perner A, Plunkett CM, Ranieri M, Schorr CA, Seckel MA, Seymour CW, Shieh L, Shukri KA, Simpson SQ, Singer M, Thompson BT, Townsend SR, Van der Poll T, Vincent JL, Wiersinga WJ, Zimmerman JL, Dellinger RP. Surviving Sepsis Campaign: International Guidelines for Management of Sepsis and Septic Shock: 2016. Intensive Care Med. 2017 Mar;43(3):304-377. doi: 10.1007/s00134-017-4683-6. Epub 2017 Jan 18. PMID 28101605
- [Background] Aspide R, Bertolini G, Albini Riccioli L, Mazzatenta D, Palandri G, Biasucci DG. A Proposal for a New Protocol for Sonographic Assessment of the Optic Nerve Sheath Diameter: The CLOSED Protocol. Neurocrit Care. 2020 Feb;32(1):327-332. doi: 10.1007/s12028-019-00853-x. PMID 31583527
- [Background] Wijdicks EF, Bamlet WR, Maramattom BV, Manno EM, McClelland RL. Validation of a new coma scale: The FOUR score. Ann Neurol. 2005 Oct;58(4):585-93. doi: 10.1002/ana.20611. PMID 16178024
- [Background] Gaastra B, Ren D, Alexander S, Awad IA, Blackburn S, Dore S, Hanley D, Nyquist P, Bulters D, Galea I. Evidence-based interconversion of the Glasgow Outcome and modified Rankin scales: pitfalls and best practices. J Stroke Cerebrovasc Dis. 2022 Dec;31(12):106845. doi: 10.1016/j.jstrokecerebrovasdis.2022.106845. Epub 2022 Oct 26. PMID 36309002
- [Background] Anderson CS, Heeley E, Huang Y, Wang J, Stapf C, Delcourt C, Lindley R, Robinson T, Lavados P, Neal B, Hata J, Arima H, Parsons M, Li Y, Wang J, Heritier S, Li Q, Woodward M, Simes RJ, Davis SM, Chalmers J; INTERACT2 Investigators. Rapid blood-pressure lowering in patients with acute intracerebral hemorrhage. N Engl J Med. 2013 Jun 20;368(25):2355-65. doi: 10.1056/NEJMoa1214609. Epub 2013 May 29. PMID 23713578